CLINICAL TRIAL: NCT04653506
Title: Non - Opioid Treatments (Single Administration) for Pain During the Early Postpartum Period After Vaginal Delivery
Brief Title: Paracetamol / Ibuprofen for Postpartum Pain in the Early Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Shmuel Kivity, MD, director head of clinical trails department, principal investigator, clinical professor, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0368-20-TLV
Record Dates: First submitted 2020-11-22; First posted 2020-12-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain
Keywords: Post Partum Pain, Pain Relief, Non-Opioids Analgesia
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: * Women participating in the study will receive postpartum analgesia immediately while reporting pain requiring analgesia (NRS <3)
  * Pain Reliefs will be given in a double-blind mechanism, in closed envelopes
  * The envelopes will contain Paracetamol 1000 mg or Ibuprofen 400 mg
  * Women participating in the study will answer a questionnaire to characterize the pain while taking the pain relief (time 0), an hour later (time 1), 4 and 6 hours later (time 4 and time 6)
Who Masked: Participant, Care Provider
Masking Description: The primary investigator will be the only one to have the information about envelopes contain
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol group (Experimental): Women who were treated with a double-blind mechanism in an envelope containing paracetamol pills (1000 mg)
  Interventions: Drug: Paracetamol 1000 mg
- Ibuprofen group (Experimental): Women who were treated with a double-blind mechanism in an envelope containing Ibuprofen pills (400 mg)
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Paracetamol 1000 mg — Women participating in the study will receive postpartum analgesia immediately while reporting pain requiring analgesia, by envelope contains paracetamol 1000 mg or ibuprofen 400 mg
  Arms: Paracetamol group
Drug: Ibuprofen 400 mg — Women participating in the study will receive postpartum analgesia immediately while reporting pain requiring analgesia, by envelope contains paracetamol 1000 mg or ibuprofen 400 mg
  Arms: Ibuprofen group

SUMMARY:
The investigators will examine the effectiveness of non-opioid analgesia (Paracetamol versus Ibuprofen) in the early postpartum period

DETAILED DESCRIPTION:
Postpartum pain is a common problem that leads to difficulties in basic daily activities, overuse of opioid medications, and even impaired breastfeeding ability. Non-opioid analgesia may play an essential role in reducing pain and improving the postpartum period including the ability to breastfeed and caring for the newborn.

This study will compare non-opioid treatment - 1000 mg Paracetamol versus 400 mg Ibuprofen in order to determine the optimal pain relief treatment in the early postpartum period that may decrease the use of opioid analgesia.

The investigators will evaluate the pain by the Numerical Rating Scale (NRS) index in the early postpartum period. The evaluation will conduct at 4-time points - while the women taking the pain relief (time 0), an hour later (time 1), 4, and 6 hours later (time 4 and time 6).

The investigators will compare the analgetic effect of each drug and evaluate the need for additional analgesia whether opioid or not.

Furthermore, the investigators will examine when women sought pain relief and whether pain relief contributes to the ability of Breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-50, who gave birth in a vaginal birth

Exclusion Criteria:

* Sensitivity to Paracetamol or Ibuprofen
* After cesarean section
* Received analgesia prior to study recruitment
* Perineal tears grade 3 \ 4
* Women with chronic pain, rheumatic disease, fibromyalgia, or trauma
* Women with a diagnosis or medication for anxiety or depression
* Dropout for women whose newborns needed respiratory support with intubation, cooling, prolonged hospitalization in NICU exceeding one week

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 107 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Pain relief after treatment with Paracetamol or Ibuprofen | 6 hours after intervention
  After getting a pain relief treatment, the participants will answer a questionnaire about pain relief at 4 - time points: the time of getting the pain relief treatment (time 0), after an hour (time 1), 4 hours (time 4), and six hours (time 6). The pain rating will be on the Numeric Rating Scale (NRS) that labeled from zero (no pain) to ten ((worst pain).

SECONDARY OUTCOMES:
Maximum pain location | 6 hours after intervention
  After getting a pain relief treatment, the participants will answer a questionnaire about pain relief at 4 - time points: the time of getting the pain relief treatment (time 0), after an hour (time 1), 4 hours (time 4), and six hours (time 6). The questionnaire will describe the maximal pain location area and the effectiveness of analgesic treatment in this area (by rating the pain on the NRS). The questionnaire will be at the time of taking the pain relief treatment (time 0), after an hour (time 1), 4 hours (time 4), and six hours (time 6)

OTHER OUTCOMES:
Effect on breastfeeding | 6 hours after intervention
  The participants will answer a questionnaire that will describe the effect of' pain relief on a woman's ability to breastfeed. The questionnaire will ask their desire to breastfeed before giving birth, did they really manage to breastfeed, and when they started breastfeeding. The investigator will describe if there is a correlation between pain relief and the ability to breastfeed.

CONTACTS AND LOCATIONS:
Overall Officials: shai ram, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Fahey JO. Best Practices in Management of Postpartum Pain. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):126-136. doi: 10.1097/JPN.0000000000000241. PMID 28277399
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Peahl AF, Dalton VK, Montgomery JR, Lai YL, Hu HM, Waljee JF. Rates of New Persistent Opioid Use After Vaginal or Cesarean Birth Among US Women. JAMA Netw Open. 2019 Jul 3;2(7):e197863. doi: 10.1001/jamanetworkopen.2019.7863. PMID 31348508
- [Background] Deussen AR, Ashwood P, Martis R. Analgesia for relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2011 May 11;(5):CD004908. doi: 10.1002/14651858.CD004908.pub2. PMID 21563142
- [Background] Wuytack F, Smith V, Cleary BJ. Oral non-steroidal anti-inflammatory drugs (single dose) for perineal pain in the early postpartum period. Cochrane Database Syst Rev. 2016 Jul 14;7(7):CD011352. doi: 10.1002/14651858.CD011352.pub2. PMID 27412362
- [Background] Davies NM. Clinical pharmacokinetics of ibuprofen. The first 30 years. Clin Pharmacokinet. 1998 Feb;34(2):101-54. doi: 10.2165/00003088-199834020-00002. PMID 9515184
- [Background] Chou D, Abalos E, Gyte GM, Gulmezoglu AM. Paracetamol/acetaminophen (single administration) for perineal pain in the early postpartum period. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD008407. doi: 10.1002/14651858.CD008407.pub2. PMID 23440827
- [Derived] Ram S, Madar D, Ram HS, Peleg G, Lior Y, Greenfeld A, Yakov G, Yogev Y, Maslovitz S. Paracetamol versus ibuprofen for early postpartum pain control: a randomized controlled trial. Arch Gynecol Obstet. 2025 Jul;312(1):51-57. doi: 10.1007/s00404-024-07797-4. Epub 2024 Nov 5. PMID 39499309